CLINICAL TRIAL: NCT06063473
Title: A Multi-center, Double-blind, Randomized, Placebo Controlled, Parallel-group Study, Comparing Trifarotene Cream 0.005% (Taro Pharmaceuticals U.S.A, Inc.) and to AKLIEF® Cream (Trifarotene 0.005%,Galderma) and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing Trifarotene Cream 0.005% to AKLIEF® Cream in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRFC-2208
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Trifarotene Cream 0.005% (Experimental): The study medication will be applied topically once daily at bedtime to the affected areas of the face as a thin layer, avoiding contact with the mouth, eyes, and other mucous membranes, for 84 consecutive days.
  Interventions: Drug: Trifarotene Cream 0.005%
- AKLIEF® Cream (Trifarotene 0.005%, Galderma Laboratories) (Active Comparator): The study medication will be applied topically once daily at bedtime to the affected areas of the face as a thin layer, avoiding contact with the mouth, eyes, and other mucous membranes, for 84 consecutive days.
  Interventions: Drug: AKLIEF® Cream (Trifarotene 0.005%, Galderma Laboratories)
- Placebo Control (Placebo Comparator): The study medication will be applied topically once daily at bedtime to the affected areas of the face as a thin layer, avoiding contact with the mouth, eyes, and other mucous membranes, for 84 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trifarotene Cream 0.005% — The study medication will be self-applied topically, on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days
  Other Names: Test Product
  Arms: Trifarotene Cream 0.005%
Drug: Placebo — The study medication will be self-applied topically, on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days
  Other Names: Vehicle
  Arms: Placebo Control
Drug: AKLIEF® Cream (Trifarotene 0.005%, Galderma Laboratories) — The study medication will be self-applied topically, on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days
  Other Names: Reference Product
  Arms: AKLIEF® Cream (Trifarotene 0.005%, Galderma Laboratories)

SUMMARY:
To demonstrate therapeutic equivalence and safety of Trifarotene cream 0.005% (Taro Pharmaceuticals U.S.A., Inc.) and AKLIEF® cream in the treatment of acne vulgaris

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, placebo-controlled, parallel-group study, comparing Trifarotene Cream 0.005% (Taro Pharmaceuticals U.S.A., Inc.) to AKLIEF® Cream and both active treatments to a placebo control in the treatment of acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Subjects who are 18 years of age or older (up to the age of 40) must have provided IRB approved written informed consent. Subjects ages 12 to 17 years of age inclusive must have provided IRB approved written assent;
* Subjects must have a definite clinical diagnosis of acne vulgaris of severity grade 2, 3,or 4 as per the Investigator's Global Assessment (IGA)
* Subjects must have ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 20 inflammatory lesions (i.e., papules and pustules) AND ≤2 nodulocystic lesions (i.e., nodules and cysts), at baseline on the face.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation
* Subjects with a history of hypersensitivity or allergy to tretinoin, retinoids, or any of the study medication ingredients.
* Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis,squamous cell carcinoma, eczema, acneiform eruptions caused by medications,steroid acne, steroid folliculitis, or bacterial folliculitis).

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 762 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Demonstration in Therapeutic Equivalence & Safety of the Investigational Product | Baseline to Week 12
  Percent change in the inflammatory (papules and pustules) & non-inflammatory (open and closed comedones) lesion counts

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals, Inc.
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No